CLINICAL TRIAL: NCT05520268
Title: Efficacy of Music Therapy and Digital Music Rehabilitation in Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other); City of Helsinki (Other)
Responsible Party: Principal Investigator, Teppo Sarkamo, Associate Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 346211; 338448 (Other Grant/Funding Number: Academy of Finland); 803466 (Other Grant/Funding Number: European Research Council)
Record Dates: First submitted 2022-08-23; First posted 2022-08-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Dementia
Keywords: music therapy; music-based rehabilitation; digital intervention; cognitive functioning; memory; emotion; mood; quality of life; electroencephalography; magnetic resonance imaging
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional music therapy (CMT) (Experimental): Participants receive 10 weeks of CMT and standard care.
  Interventions: Behavioral: Conventional music therapy (CMT)
- Digital music rehabilitation (DMR) (Experimental): Participants receive 10 weeks of DMR and standard care.
  Interventions: Behavioral: Digital music rehabilitation (DMR)
- Standard care (No Intervention): Participants receive only standard care. Standard care comprises normal care services received by the PWDs in the Finnish health care system.

INTERVENTIONS:
Behavioral: Conventional music therapy (CMT) — CMT comprises both receptive and expressive musical activities (listening and reminiscing to music, singing, and moving to music) held in small groups (8 PWDs/group) for a duration of 10 weeks (2x60 min sessions/week) and led by a professional music therapist. For PWDs living in a care home, the CMT sessions are implemented as inpatient rehabilitation held at the care home. For PWDs living at home, the CMT sessions are implemented as outpatient rehabilitation held at a local day activity centre.
  Arms: Conventional music therapy (CMT)
Behavioral: Digital music rehabilitation (DMR) — DMR comprises both receptive and expressive musical activities (listening and reminiscing to music, singing, and moving to music) held in small groups (8 PWDs/group) for a duration of 10 weeks (2x60 min sessions/week) and implemented using a novel digital music content service called HILDA. In HILDA, there are a number of stand-alone musical programs hosted by a virtual presenter which the PWDs can follow and through which they can interact. The DMR sessions are moderated by an instructor (care home staff member or research assistant). For PWDs living in a care home, the DMR is implemented as live sessions held at the care home using a HILDA box connected to a TV screen and operated via a remote controller by the instructor. For PWDs living at home, the DMR is implemented as virtual sessions using a video communication platform that allows the instructor to stream and control the HILDA service and the participants to see and hear each other and interact.
  Arms: Digital music rehabilitation (DMR)

SUMMARY:
This study evaluates the applicability and clinical efficacy of conventional music therapy and digital music rehabilitation for dementia in home and care home settings.

DETAILED DESCRIPTION:
Rationale: In persons with dementia (PWDs), music-based interventions have shown positive effects on emotional, behavioural and cognitive symptoms as well as on psychological well-being and quality of life. Despite the evidence for the efficacy of music in PWDs, many issues surround the practicalities of music interventions, especially regarding their applicability, scalability, and optimization across the dementia care continuum. Moreover, the individual factors affecting the treatment outcomes of music-based interventions remain largely unexplored in dementia.

Aims: The purpose of this randomized controlled trial (RCT) is to determine the applicability and clinical efficacy of conventional music therapy and digital music rehabilitation for dementia in both home and care home settings. Specifically, the RCT seeks to determine (i) can conventional music therapy (CMT) and digital music rehabilitation (DMR) enhance or support cognitive function, mood, and quality of life in dementia compared to standard care; (ii) how does the efficacy of CMT and DMR differ in the different stages of dementia; and (iii) how do baseline demographic factors (e.g., age, gender, education), musical factors (musical background, music cognition) and neural factors (e.g., extent of neuropathology, preservation of music networks) affect the efficacy of the music interventions.

Methods: Participants are 192 PWDs across the dementia care continuum (PWDs with mild-moderate dementia living at home and PWDs with moderate-severe dementia living in care homes; N=96 each). Following a three-arm parallel-group RCT design, the PWDs living at home and at care homes are randomized into three groups (CMT, DMR, standard care; N=32 each]. The CMT and DMR comprise passive and active engagement with music over 10 weeks (2x60 min sessions/week), implemented either by a music therapist (CMT) or using a novel digital music content service (DMR). To investigate the efficacy of the music interventions, participants complete measures of cognitive functioning (neuropsychological tests) and mood and quality of life (questionnaires, clinical scales), which are assessed at three time points: baseline (pre-intervention), 3-month stage (post-intervention) and 6-month stage (follow-up). Additionally, family member and caregivers of PWDs are asked to answer questionnaires on the psychological well-being of the PWD (informant-report) and themselves (self-report). To explore the individual musical and neural factors that may affect the efficacy of music interventions, participants also complete a musical assessment battery as well as electroencephalography (EEG) and structural and functional MRI (s/fMRI) measurements at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed dementia (according to International Classification of Diseases [ICD] criteria), which is mild [Clinical Dementia Rating (CDR) score: 0.5-1, Global Deterioration Scale (GDS) score: 3-4], moderate (CDR: 2, GDS: 4-6), or severe (CDR: 3, GDS: 6-7) dementia
* Age ≥ 60 years
* Finnish-speaking (or bilingual; the study is performed in Finnish)
* Stable physical and somatic condition (no major changes in psychotropic medication during the last 3 months)
* Physically and cognitively able to take part in the intervention and assessments.

Exclusion Criteria:

* Prior severe psychiatric illness or substance abuse
* Major hearing or visual impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the MoCA score at 3-month stage | Baseline and 3-month stage
  Montreal Cognitive Assessment (MoCA) score (range 0-30, higher score indicates better outcome), measures general cognitive function
Change from baseline in the CERAD total score at 3-month stage | Baseline and 3-month stage
  Consortium to Establish a Registry for Alzheimer's Disease (CERAD) total score (Chandler score, range 0-100, higher score indicates better outcome), measures general cognitive function

SECONDARY OUTCOMES:
Change from baseline in the MoCA score at 6-month stage | Baseline and 6-month stage
  Montreal Cognitive Assessment (MoCA) score (range 0-30, higher score indicates better outcome), measures general cognitive function
Change from baseline in the CERAD total score at 6-month stage | Baseline and 6-month stage
  Consortium to Establish a Registry for Alzheimer's Disease (CERAD) total score (Chandler score, range 0-100, higher score indicates better outcome), measures general cognitive function
Change from baseline in the MoCA Fluency score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Montreal Cognitive Assessment (MoCA) Fluency subtest score (phonemic fluency; min: 0, max: no upper limit, higher score indicates better outcome), measures language skills
Change from baseline in the CERAD Fluency score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Fluency subtest score (semantic fluency; min: 0, max: no upper limit, higher score indicates better outcome), measures language skills
Change from baseline in the CERAD Naming score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Naming subtest score (range: 0-15, higher score indicates better outcome), measures language skills
Change from baseline in the CERAD Constructional Praxis score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Constructional Praxis subtest score (range: 0-11, higher score indicates better outcome), measures visuoconstructive function
Change from baseline in the CERAD Word List Learning score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Word List Learning subtest score (range: 0-30, higher score indicates better outcome), measures verbal learning
Change from baseline in the CERAD Word List Recall score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Word List Recall subtest score (range: 0-10, higher score indicates better outcome), measures delayed spontaneous verbal recall
Change from baseline in the CERAD Word List Recognition score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Word List Recognition subtest score (range: 0-20, higher score indicates better outcome), measures delayed cued verbal recall
Change from baseline in the WMS-IV Logical Memory I score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Wechsler Memory Scale IV (WMS-IV) Logical Memory I subtest score (range: 0-56, higher score indicates better outcome), measures immediate verbal recall
Change from baseline in the WMS-IV Logical Memory II score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Wechsler Memory Scale IV (WMS-IV) Logical Memory II subtest score (range: 0-28, higher score indicates better outcome), measures delayed verbal recall
Change from baseline in the IFS total score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  INECO Frontal Screening (IFS) total score (range 0-30, higher score indicates better outcome), measures executive function and working memory
Change from baseline in the IFS Executive subscore at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  INECO Frontal Screening (IFS) Executive subscore (summary score of the Motor Series, Conflicting Instructions, Go-No Go, Proverbs and Hayling Test subtests, range 0-18, higher score indicates better outcome), measures executive function
Change from baseline in the IFS Working memory subscore at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  INECO Frontal Screening (IFS) Working memory subscore (summary score of the Digits Backward, Verbal Working Memory and Spatial Working Memory subtests, range 0-12, higher score indicates better outcome), measures working memory
Change from baseline in autobiographical memory score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Custom-made autobiographical memory questionnaire, percentage score (range 0-100, higher score indicates better outcome; also qualitative data collected), measures subjective and objective autobiographical memory
Change from baseline in the MADRS score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Montgomery-Åsberg Depression Rating Scale (MADRS) score (range 0-60, higher score indicates worse outcome), measures depression symptoms
Change from baseline in the PROMIS Depression score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Patient-Reported Outcomes Measurement Information System (PROMIS) Depression scale score (range 8-40, higher score indicates worse outcome), measures depression symptoms
Change from baseline in the PROMIS Anxiety score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety scale score (range 8-40, higher score indicates worse outcome), measures anxiety symptoms
Change from baseline in the NPI-Q Severity score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Neuropsychiatric Inventory Questionnaire (NPI-Q) Severity scale score (range 0-36, higher score indicates worse outcome), measures the severity of neuropsychiatric symptoms
Change from baseline in the NPI-Q Distress score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Neuropsychiatric Inventory Questionnaire (NPI-Q) Distress scale score (range 0-60, higher score indicates worse outcome), measures the distress caused by the neuropsychiatric symptoms on caregivers
Change from baseline in the NPI-Q total score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Neuropsychiatric Inventory Questionnaire (NPI-Q) total score (range 0-180, calculated as Severity x Distress, higher score indicates worse outcome), measures the total level of neuropsychiatric symptoms
Change from baseline in the QoL-AD score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Quality of Life in Alzheimer's Disease (QoL-AD) score (range 15-60, higher score indicates better outcome), measures quality of life
Change from baseline in the EuroQol EQ-5D-5L Health index score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  EuroQol EQ-5D-5L Health index score (range 0-1, higher score indicates better outcome), measures health-related quality of life
Change from baseline in the EuroQol EQ-5D-5L Health VAS score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  EuroQol EQ-5D-5L Health VAS score (range 0-100, higher score indicates better outcome), measures general health
Change from baseline in the caregiver GHQ-12 score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  General Health Questionnaire 12 (GHQ-12) score (caregiver self-report; range 0-36, higher score indicates worse outcome), measures stress and psychological well-being
Change from baseline in the caregiver ZBI-12 score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Zarit Burden Interview 12 (ZBI-12) score (caregiver self-report; range 0-48, higher score indicates worse outcome), measures caregiver burden
Change from baseline in the UWES-9 score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Utrecht Work Engagement Scale 9 (UWES-9) score (nurse self-report; range 0-54, higher score indicates better outcome), measures occupational well-being
Change from baseline in the PCTB score at 3-month and 6-month stages | Baseline, 3-month stage and 6-month stage
  Professional Care Team Burden (PCTB) score (nurse self-report; range 0-40, higher score indicates worse outcome), measures professional care team burden

OTHER OUTCOMES:
Association between baseline demographic and musical background factors and change in primary/secondary outcome measures (from baseline to 3-month and 6-month stages) | Baseline
  Demographic (e.g., age, gender, education) and musical (e.g., previous and current musical activity, music education) factors at baseline (data collected using interview / questionnaires). These data are used as predictors of treatment effects in the primary/secondary outcome measures.
Association between baseline music cognition indices and change in primary/secondary outcome measures (from baseline to 3-month and 6-month stages) | Baseline
  Different elements of music cognition (music perception, musical emotions, rhythmic timing, musical movement, singing) measured at baseline using questionnaires and short behavioural tasks. These data are used as predictors of treatment effects in the primary/secondary outcome measures.
Association between baseline ERP indices and change in primary/secondary outcome measures (from baseline to 3-month and 6-month stages) | Baseline
  Amplitude and latency of event-related potentials (ERPs) linked to auditory perception and memory in two passive auditory tasks measured at baseline using electroencephalography (EEG). These data are used as predictors of treatment effects in the primary/secondary outcome measures.
Association between baseline sMRI indices and change in primary/secondary outcome measures (from baseline to 3-month and 6-month stages) | Baseline
  Grey matter volume in cortical and subcortical brain regions measured at baseline using structural magnetic resonance imaging (sMRI: MPRAGE sequence). These data are used as predictors of treatment effects in the primary/secondary outcome measures.
Association between baseline dMRI indices and change in primary/secondary outcome measures (from baseline to 3-month and 6-month stages) | Baseline
  Structural connectivity of white matter tracts measured at baseline using diffusion magnetic resonance imaging (dMRI: HARDI sequence). These data are used as predictors of treatment effects in the primary/secondary outcome measures.
Association between baseline fMRI indices and change in primary/secondary outcome measures (from baseline to 3-month and 6-month stages) | Baseline
  Brain activation and connectivity at resting state and during music listening measured at baseline using functional magnetic resonance imaging (fMRI). These data are used as predictors of treatment effects in the primary/secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Teppo Särkämö, PhD, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki / Faculty of Medicine / Department of Psychology, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in articles, after deidentification
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.